CLINICAL TRIAL: NCT03731702
Title: Optimization of Collection Methods for Studies of the Human Microbiota
Status: Withdrawn | Type: Observational
Why Stopped: Deemed not human subjects research
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919013; 19-C-N013
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Microbial Composition
Keywords: Oral Microbiota; Fecal Microbiota; Stability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- General Individuals: Any adult working at the NCI who has not used antibiotics in the past 3 months.

SUMMARY:
Background:

The human microbiota is the bacteria and other microbes found in and on the human body. Scientists study the microbiota because it is related to many health conditions. The way samples are collected and handled can greatly affect microbiota study findings. Researchers want to learn more about how collection methods affect these studies.

Objectives:

To compare different oral and fecal collection methods. To test the effect of new methods to get DNA out of these samples.

Eligibility:

Adults ages 18 and older who are National Cancer Institute employees and have not taken antibiotics in the past 3 months

Design:

Participants will discuss the study with researchers.

Participants will give an oral or fecal sample or both.

For the oral sample, participants will be told what not to do beforehand. This includes chewing gum and smoking. Participants will spit saliva into a tube. Then they will get mouthwash in a vial. They will swish and gargle the mouthwash for 30 seconds then spit it back in the vial.

Participants giving a fecal sample will get a collection kit. They can collect the sample at home or elsewhere. Participants will have a bowel movement into the collection container. They will smear some of it on a card with a stick and put the rest in 2 tubes. They will mix the feces with the solution in the tubes. Participants will write the date and time of collection on the instructions and return the sample within 24 hours.

Participants providing both samples could have 3 study visits: 1 to give an oral sample, 1 to get the fecal sample collection kit, and 1 to return that sample.

DETAILED DESCRIPTION:
The human microbiome (i.e., the collection of microbial genes found in and on the human body) has been observed to be associated with numerous health conditions, but current methodological studies suggest that collection method, laboratory handling, bioinformatic processing of the data, and other factors can greatly affect microbiome study findings. In cohort studies, samples should be collected using validated methods that can be analyzed using multiple technologies, however these technologies and methods are regularly changing and being modified. Therefore, we need to test multiple collection methods for new technologies or test new collection methods to assess the comparability of the results. We will evaluate the effect of several collection methods for oral and/or fecal samples from 100 individuals who work at the NCI on microbial characteristics. Once the samples are collected, we will create aliquots and store the samples for further processing. We will then test the effect of new DNA extraction methods, sequencing technologies, and bioinformatics pipelines using these samples. Any remaining aliquots will remain in the -80 degrees Celsius freezer for other future studies. This study will be essential to understand the impact of collection methods for oral and fecal samples for future epidemiologic studies.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Adults who work at the NCI, either in Shady Grove or in the Advanced Technology Center (ATC)
* Willing to provide oral and/or fecal samples.
* At least 18 years of age or older
* Not taken antibiotics anytime in the past 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit 100 adults who work at the NCI, either in Shady Grove or in the Advanced Technology Center (ATC), who are willing to provide oral and/or fecal samples. We will include any participant that is at least 18 years of age or older who is employed at NCI and has not taken antibiotics anytime in the past 3 months since antibiotic use has been shown to disrupt the microbiota.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Oral and/or fecal microbiota | 1 month
  relative abundance and phylogenetic diversity of their oral and/or fecal microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Vogtmann, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- NIH NCI Shady Grove, Rockville, Maryland, United States